CLINICAL TRIAL: NCT00822224
Title: Use of MEOPA for Elderly With Dementia.
Brief Title: Use of MEOPA (Equimolar Mixture of Nitrogen Protoxide and Oxygen) for Elderly With Dementia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Collaborators: Fondation de France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08-PP-03
Record Dates: First submitted 2009-01-13; First posted 2009-01-14 (Estimated); Last update posted 2011-12-09 (Estimated); Status verified 2011-12

CONDITIONS: Dementia
Keywords: acute pain; MEOPA; Dementia
MeSH Terms: conditions — Dementia; Acute Pain | interventions — Meopa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Use of MEOPA during the painful care
  Interventions: Drug: MEOPA

INTERVENTIONS:
Drug: MEOPA — inhalation of MEOPA during the painful care

SUMMARY:
Acute pain is frequent in elderly especially in geriatrics acute care units where painful procedures are often occurring.

MEOPA represents an alternative to opioïd therapy to prevent procedural pain during the treatment of pressure ulcers.

In this study, cognitive impairment and dementia do not limit the use of MEOPA. The new approach in the management of acute procedural pain provides effective and safe analgesia in frail old patients.

ELIGIBILITY:
Inclusion Criteria:

* dementia (Folstein scoring between 0 and 25)
* older than 75
* health necessitating of painful care for example eschar care

Exclusion Criteria:

* bullous emphysema
* pneumothorax

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2009-01; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
feasibility of use of MEOPA as tolerance to mask, MEOPA inhalation | one time, at the first care with MEOPA

SECONDARY OUTCOMES:
satisfaction rate of patient | one time, at the first care with MEOPA

CONTACTS AND LOCATIONS:
Overall Officials: Françoise CAPRIZ-RIBIERE, PhD, Principal Investigator — Gerontology department, Nice University Hospital
Locations (1):
- Gerontology department, Nice University Hospital, Nice, France